CLINICAL TRIAL: NCT06255366
Title: Analysis of the Clinical Efficacy of Intravenous Application of Hemostatic Drugs in Improving the Clarity of Vision Under Endoscope, Perioperative Bleeding Volume and Anti-inflammatory Effect of Spinal Endoscopic Lumbar Fusion
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Chengdu University of Traditional Chinese Medicine (Other)
Responsible Party: Principal Investigator, Fei Yang, Deputy director, Chengdu University of Traditional Chinese Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2023KL-138
Record Dates: First submitted 2024-01-23; First posted 2024-02-13 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: Lumbar Spondylolisthesis; Arthrosis; Spine
Keywords: Lumbar Spondylolisthesis; Carbazochrome; Desmopressin; Endoscope
MeSH Terms: conditions — Spondylolisthesis; Osteoarthritis | interventions — Deamino Arginine Vasopressin; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Caroxime sodium sulfonate (Experimental): Five minutes before surgery, intravenous infusion of caroxime sodium sulfonate and sodium chloride injection 100ml (80mg) (trade name: Weiluojing, 100ml, containing caroxime sodium sulfonate 80mg and sodium chloride 0.9g, Chongqing Dikang Changjiang Pharmaceutical Co., LTD.) was given, and intravenous infusion of caroxime sodium sulfonate and sodium chloride injection 100ml (80mg) was given again 1 hour after surgery.
  Interventions: Drug: Caroxime sodium sulfonate
- Desmopressin (Experimental): Intravenous infusion of desmopressin injection 4ug (Shenzhen Hanyu) +0.9% sodium chloride injection 100ml was given 5 minutes before surgery, and intravenous infusion of desmopressin injection 4ug (Shenzhen Hanyu) +0.9% sodium chloride injection 100ml was given again 1 hour after surgery
  Interventions: Drug: Desmopressin
- 0.9% Sodium chloride injection (Placebo Comparator): Intravenous infusion of 0.9% sodium chloride injection 100ml (specification 100ml, containing 0.9g sodium chloride, Sichuan Kelun Pharmaceutical Co., LTD.) was given 5 minutes before surgery, and intravenous infusion of 0.9% sodium chloride injection 100ml was given again 1 hour after surgery
  Interventions: Drug: 0.9% Sodium Chloride Injection

INTERVENTIONS:
Drug: Caroxime sodium sulfonate — Five minutes before surgery, intravenous infusion of caroxime sodium sulfonate and sodium chloride injection 100ml (80mg) (trade name: Weiluojing, 100ml, containing caroxime sodium sulfonate 80mg and sodium chloride 0.9g, Chongqing Dikang Changjiang Pharmaceutical Co., LTD.) was given, and intravenous infusion of caroxime sodium sulfonate and sodium chloride injection 100ml (80mg) was given again 1 hour after surgery.
  Arms: Caroxime sodium sulfonate
Drug: Desmopressin — Intravenous infusion of desmopressin injection 4ug (Shenzhen Hanyu) +0.9% sodium chloride injection 100ml was given 5 minutes before surgery, and intravenous infusion of desmopressin injection 4ug (Shenzhen Hanyu) +0.9% sodium chloride injection 100ml was given again 1 hour after surgery
  Arms: Desmopressin
Drug: 0.9% Sodium Chloride Injection — Intravenous infusion of 0.9% sodium chloride injection 100ml (specification 100ml, containing 0.9g sodium chloride, Sichuan Kelun Pharmaceutical Co., LTD.) was given 5 minutes before surgery, and intravenous infusion of 0.9% sodium chloride injection 100ml was given again 1 hour after surgery
  Arms: 0.9% Sodium chloride injection

SUMMARY:
To study the clinical efficacy of carosodiumsulfonate and desmopressin in improving the clarity of vision under endoscope, perioperative bleeding volume and anti-inflammatory effect in endoscopic lumbar fusion

DETAILED DESCRIPTION:
A total of 129 patients diagnosed with lumbar spondylolisthesis and undergoing endoscopic lumbar fusion in our hospital from February 2024 to February 2025 were prospectively enrolled in this trial. All subjects who met the inclusion criteria were enrolled in the trial after signing the informed consent form. After completing the relevant information registration, routine preoperative preparation was performed and relevant baseline data were collected. The randomization scheme was completed by specialized statisticians independently and was not affected by the subjective will of the researchers and the subjects. According to the random number table method, all subjects were equally allocated to group A, group B and group C at a ratio of 1:1:1. Participants and investigators were blinded to group assignments until the end of the study and were blinded only if a participant developed a serious complication during treatment. Blood routine, liver function, renal function, electrolytes, coagulation indexes and other hematological tests were routinely performed before operation. The volume of blood drawn was about 15ml. Experimental group (group A) : Intravenous infusion of caroxime sodium sulfonate and sodium chloride injection 100ml (caroxime sodium sulfonate 80mg and sodium chloride 0.9g) (Chongqing Dikang) was given 5 minutes before operation. One hour after operation, intravenous infusion of carosene sodium sulfonate injection 100ml (carosene sodium sulfonate 80mg and sodium chloride 0.9g) (Chongqing Dicang) [reference to Weiluojing (Carosene sodium sulfonate sodium chloride injection) 100ml (80mg: 0.9g) Usage and dosage: intravenous infusion of 80mg each time (approval number: Chinese Medicine approval number H20052472)]; Experimental group (group B) : Intravenous infusion of desmopressin injection 15ug (Shenzhen Hanyu) +0.9% sodium chloride injection 100ml 5 minutes before surgery, intravenous infusion of desmopressin injection 15ug (Shenzhen Hanyu) +0.9% sodium chloride injection 100ml 1 hour after surgery [according to the instructions of desmopressin injection (Hangu), usage and dosage: 1. Control of bleeding or prevention of bleeding before operation: according to the dose of 0.3ug/kg body weight, diluted to 50-100ml with normal saline, intravenous infusion within 15-30min (approval number: H20064093); In control group (group C), 100ml 0.9% sodium chloride solution was intravenously infused 5 minutes before surgery and again 1 hour after surgery. Intraoperative Gertzbein-Sload (GS) score was used to score the clarity of the intraoperative visual field under the microscope. During the operation, the operation time and the total amount of perfusate were recorded, and the red blood cell count was measured by taking the perfusate from the drainage bottle. The blood routine, erythrocyte sedimentation rate, CRP and IL-6 were rechecked at 3 days, and the amount of blood drawn was about 10ml each time. The total blood loss, intraoperative blood loss and hidden blood loss of the patients were recorded, and the VAS scores at 1 day, 2 days and 3 days after operation were recorded. To evaluate the effect of intravenous administration of carosodiumsulfonate and desmopressin on the clarity of visual field under endoscope, perioperative blood loss and postoperative inflammatory indicators in endoscopic lumbar fusion.

ELIGIBILITY:
Inclusion Criteria:

1. Patients, aged 35-65 years old, who were diagnosed as single-segment lumbar spondylolisthesis without spondylolysis based on imaging data and underwent endoscopic lumbar interbody fusion.
2. In patients with normal platelet count, blood coagulation function.
3. No history of major lumbar trauma and previous lumbar surgery.
4. No allergy history, contraindications and serious adverse reactions to desmopressin and carosodiumsulfonate.
5. American Society of Anesthesiologists (ASA) classification: grade 1-2
6. The participants and their family members were informed of the nature of the study, understood the provisions of the study, complied well, and signed informed consent

Exclusion Criteria:

1. Patients who do not consent to participate in the trial.
2. Poorly controlled hypertension with systolic blood pressure >180 mmHg or diastolic blood pressure >110 mmHg.
3. People with mental illness, or poor compliance of patients.
4. Patients with severe liver function impairment and creatinine clearance <20ml/min.
5. Patients with coagulopathy or inability to tolerate surgery.
6. Patients with other lumbar spine diseases or pulmonary tuberculosis.
7. ASA anesthesia level 3 or higher.
8. Patients with a long history of smoking, alcohol abuse, or contraceptive drug abuse.
9. Patients with serious heart disease, diabetes.
10. Imaging tip is merged with other lumbar disease or accompanied by lumbar spondylolysis patients.
11. Pregnant women.
12. Patients with a history of major lumbar trauma or lumbar surgery.

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Estimated)
Dates: Start 2024-03-28 (Estimated); Primary Completion 2024-12-30 (Estimated); Study Completion 2025-06-29 (Estimated)

PRIMARY OUTCOMES:
Clarity under microscope | During the operation
  Grade 1: Vital areas cannot be seen clearly but is sufficient to perform surgery. Means that the visual field quality of the operation is low, but sufficient for simple surgical procedures. Grade 2: Visual field clarity is good enough to perform fast and accurate surgery. It means that the quality of the surgical field is good and the operation can be performed efficiently. Grade 3: Excellent visual acuity, can perform difficult surgery. It means that the surgical field is very clear and can perform difficult operations.
Total Blood Loss（TBL） | During the operation
  Preoperative blood volume was calculated according to the Nadler equation, preoperative blood volume (PBV)=K1× height (m)3+ K2× body weight (kg) + K3(male: K1=0.366 9, K2=0.032 19, K3=0.604 1; Female: K1=0.356 1, K2=0.033 08, K3=0.183 3). The Delphi formula was used to calculate the total blood loss of patients, total blood loss = preoperative blood volume ×2× (preoperative hematocrit - postoperative hematocrit)/(preoperative hematocrit + postoperative hematocrit)
Intraoperative Blood Loss（IBL） | During the operation
  Intraoperative Blood Loss (IBL) : IBL = Amount of fluid collected from the drainage bottle + Weight increase of gauze used during the operation - Amount of lavage fluid used during the operation
Hidden Blood Loss（HBL） | During the operation
  Hidden Blood Loss（HBL） = Total Blood Loss（TBL） -Intraoperative Blood Loss（IBL）
Duration of surgery | During the operation
Intraoperative perfusion fluid consumption | During the operation
Red blood cells were counted in the postoperative drainage fluid | Up to 72 hours after surgery
Intraoperative blood pressure values | During the operation
  Systolic and diastolic blood pressure

SECONDARY OUTCOMES:
Erythrocyte sedimentation Rate（ESR） | Up to 72 hours after surgery
Visual analogue scale | Up to 72 hours after surgery
  Pain was evaluated using a visual analogue scale (VAS) where 0 was no pain and 10 was unbearable pain.
IL--6 | Up to 72 hours after surgery
  Interleukin- 6
C-reactive protein | Up to 72 hours after surgery